CLINICAL TRIAL: NCT06405776
Title: Effect of Perioperative Continuous Intravenous Infusion of Lidocaine on Postoperative Pain and Long-term Survival in Elderly Patients Undergoing Colorectal Cancer Surgery: a Prospective, Randomized Controlled Trial
Brief Title: Effect of Lidocaine on Postoperative Pain and Long-term Survival in Elderly Patients Undergoing Colorectal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: West China Hospital (Other)
Responsible Party: Principal Investigator, Chunling Jiang, Professor, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2020HX1180-2
Record Dates: First submitted 2024-05-05; First posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine group (Experimental): Patients in the lidocaine group, lidocaine 1.5mg/kg/h is continuously infused (using ideal body weight) during the whole procedure, postoperative analgesia pump with lidocaine (lidocaine 50mg/kg, sufentanil 2ug/kg, glassetron 12mg) diluted to 200ml with saline until 72h after surgery.
  Interventions: Drug: lidocaine
- Placebo group (Placebo Comparator): In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2μg/kg, granisetron 12mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 mL.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: lidocaine — Patients in the lidocaine group, lidocaine 1.5mg/kg/h is continuously infused (using ideal body weight) during the whole procedure, postoperative analgesia pump with lidocaine (lidocaine 50mg/kg, sufentanil 2ug/kg, glassetron 12mg) diluted to 200ml with saline until 72h after surgery.
  Arms: Lidocaine group
Drug: Placebo — In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2μg/kg, granisetron 12mg diluted to 200 mL in 0.9% normal saline solution with a total volume of 200 mL.
  Arms: Placebo group

SUMMARY:
This study is a further observation and follow-up of the patients enrolled in the registration number NCT05920980 to further evaluate the effect of long-term infusion of lidocaine on postoperative chronic pain, long-term quality of life and survival rate in patients undergoing colorectal cancer surgery.

DETAILED DESCRIPTION:
This study is a further observation and follow-up of the patients enrolled in the registration number NCT05920980 to further evaluate the effect of long-term infusion of lidocaine on postoperative chronic pain, long-term quality of life and survival rate in patients undergoing colorectal cancer surgery. Patients who meet the enrollment criteria will be randomized 1:1 to the lidocaine group or placebo group. In the lidocaine group, lidocaine 1.5mg/kg/h was continuously infused (using ideal body weight) during the whole procedure. Postoperative analgesia pump with lidocaine (lidocaine 50mg/kg, sufentanil 2ug/kg, glassetron 12mg) diluted to 200ml with saline until 72h after surgery. In the placebo group, the same volume of normal saline will be administered during anesthesia. The postoperative PCIA device will contain sufentanil 2μg/kg, granisetron 12mg diluted to 200mL in 0.9% normal saline solution with a total volume of 200mL.Follow-up after discharge includes chronic pain, the impact of chronic pain on quality of life, the relapse-free survival and overall survival from postoperative 3 months to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants were at least 60 years old;
2. American Society of Anesthesiologists (ASA) physical status I to III;
3. Body-mass index of 18-30 kg/m2;
4. Scheduled for elective colorectal surgery.

Exclusion Criteria:

1. Metastases occurring in other distant organs;
2. Severe hepatic insufficiency (aspartate aminotransferase or alaninetransaminase or bilirubin >2.5 times the upper limit of normal);
3. Renal impairment (creatinine clearance <60 mL/min);
4. Cardiac rhythm disorders or systolic heart failure (second-and thirddegree heart block, ejection fraction <50%);
5. Allergies to any of the trial drugs; chronic opioid use;
6. Inability to comprehend numeric rating scale.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of chronic pain at 3 months postoperatively | 3 months postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain,0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience.

SECONDARY OUTCOMES:
The incidence of chronic pain at 6 months ,1 year, 3 years and 5 years postoperatively | 6 months, 1 year and 3 years postoperatively
  Chronic pain is defined as pain that lasts or recurs for longer than 3 months. For chronic postsurgical pain(CPSP), it mainly refers to the pain that persists past normal healing time. Pain scoring is performed at 3 months using the Numerical Rating Scale(NRS), with 11 digits ranging from 0 to 10 indicating the degree of pain,0 indicating no pain, and 10 indicating severe pain. Subjects choose a number to indicate the degree of pain based on their personal pain experience.
Overall survival after surgery | 6 months, 1 year, 3 years, 5 years postoperatively
  Overall survival is defined as the time between the date from surgery to the date of death.
Recurrence-free survival after surgery | 6 months, 1 year, 3 years, 5 years postoperatively
  Postoperative re-examination is based on the diagnosis of enhanced CT, MRI, ultrasound or blood examination to determine whether the patient has recurrence and metastasis. Recurrence-free time refers to the time from surgery to tumor recurrence based on the above CT, MRI, etc.
Disability-free surviva survival | 6 months, 1 year, 3 years, 5 years postoperatively
  Patient self-assessment is carried out by using the World Health Organization(WHO) Disability Scale, with a minimum score of 12 points and a maximum score of 60 points. The lower the score, the higher the quality of life.
The prevalence of neuropathic pain | 3 months, 6 months, 1 year, 3 years, 5 years postoperatively
  The ID Pain scale is used as a validated assessment of neuropathic pain. ID pain questionnaire consists of six items. Pain higher scores suggest a neuropathic component to the pain.
Brief Pain Inventory(BPI) pain interference subscale score | 3 months, 6 months, 1 year, 3 years, 5 years postoperatively
  BPI pain interference subscale is a 7-item questionnaire asking participants to describe how pain has interfered general activity, mood, walking, normal work, relations with others, sleep, and enjoyment of life. Each question is answered on a scale 0(does not interfere) to 10(completely interferes). The total range of score is 0-70. The higher the scores suggest the worse the interference.

CONTACTS AND LOCATIONS:
Overall Officials: Chunling Jiang, PhD, Study Director — West China Hospital
Locations (1):
- China, Sichuan, China

IPD SHARING:
Plan to Share IPD: No